CLINICAL TRIAL: NCT00588692
Title: Strategies for Aggressive Central Afterload Reduction in Patients With Heart Failure
Acronym: SACAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AtCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Barry Borlaug, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-002008
Record Dates: First submitted 2007-12-21; First posted 2008-01-08 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Afterload Reduction; Sphygmocor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SphygmoCor Unblinded (Active Comparator): The use of the sphygmocor values will determine medication adjustments to optimize HF treatment.
  Interventions: Device: SphygmoCor
- SphygmoCor Blinded (Placebo Comparator): Sphygmocor values will be blinded to the investigator.
  Interventions: Device: SphygmoCor

INTERVENTIONS:
Device: SphygmoCor — The SphygmoCor, a hand-held tonometer will assess central blood pressure noninvasively. This pencil-like device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure.

SUMMARY:
Heart failure (HF) is the leading cause of hospitalization among Americans over the age of 65 years, affecting greater than 5 million in the U.S. alone. Significant improvements in morbidity and mortality have been achieved through the use of medications that antagonize adverse neurohormonal signaling pathways, particularly therapies that reduce left ventricular (LV) afterload.

Vascular stiffness increases with aging, contributing to the increase in cardiac load. One important repercussion of such stiffening is an increase in pulse wave velocity. As the incident pressure wave generated by cardiac ejection encounters zones of impedance mismatch (such as arterial bifurcations), part of the wave is reflected backward, summing with the incident wave, increasing central blood pressure (CBP). With normal aging, hypertension, and heart failure, increased wave velocity causes the reflected wave to reach the heart earlier, in mid to late systole, considerably increasing late-systolic load, impairing cardiac ejection, and diastolic relaxation in the ensuing cardiac cycle.

The magnitude of this reflected pressure wave can be quantified by the augmentation index (AIx). The use of vasoactive agents which antagonize this increase in late systolic load (and AIx) may prove useful in the treatment of heart failure, by facilitating cardiac ejection during late systole when reflected pressure waves predominate. However, it has never been conclusively shown in humans that CBP-targeted therapy is useful in the management of HF.

LV afterload, measured centrally in the ascending aorta, may differ considerably from brachial cuff-measured pressure, and has traditionally required invasive hemodynamic assessment to determine, limiting the applicability of techniques targeting CBP and late-systolic load. Recently, a novel, hand-held tonometer (SphygmoCor, Atcor Medical) has been developed for the noninvasive assessment of CBP. This pencil-like device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure. This device has received FDA approval for clinical use in the assessment of central pressures. However, it remains unknown whether knowledge of CBP and late-systolic load (AIx) confers any clinically-significant incremental benefit in the management of patients with heart failure. The primary objective of the proposed investigation will be to determine if this assessment might have such a role.

DETAILED DESCRIPTION:
Research Design and Methods

Hypotheses Knowledge of central aortic pressure waveforms (central pressure therapy, CPT) will affect the intensity of antihypertensive medication prescription, and treatment decisions based upon this knowledge in turn will lead to an enhanced reduction in CBP and AIx. Finally, it is hypothesized that this reduction in AIx/CBP will lead to improved exercise performance and LV systolic and diastolic reserve function.

Basic Study Plan This is a single-blind, randomized, controlled, parallel group intervention study examining the effects of a novel, noninvasive diagnostic test for determining AIx and CBP (SphygmoCor, Atcor Medical) on medical care, blood pressure control, exercise performance, and LV functional reserve in patients with chronic heart failure (HF) and systolic dysfunction (25%<EF<50%) and with preserved systolic function (EF>50%). Eligible subjects will undergo resting echocardiogram, noninvasive CBP assessment, and metabolic exercise stress testing on a recumbent cycle ergometer to quantify exercise performance. Echocardiography and CBP assessment will be performed at rest, during graded exercise, and immediately after peak exercise to determine indexes of LV systolic and diastolic performance and changes in CBP. Subjects will then be randomized (1:1) to subsequent determination of CBP at 1 month heart failure clinic visits versus sham (tonometry information acquired, but not shared with investigator). Investigators will then make adjustments to subject's medical therapy and antihypertensive regimen based upon the additional data procured via the Sphygmocor device. Subjects randomized to sham will have adjustments made as per standard clinical judgment based upon brachial blood pressure assessment and other clinical variables. In addition to standard clinical assessment, each subject will undergo 6 minute walk test at each visit, administered by the study coordinator.

At the 6 month follow up visit, subjects will undergo resting and exercise echo/CBP/metabolic stress testing exactly as performed at visit 1. The co-primary endpoints will be the change in central augmentation index (defined below) and change in peak oxygen uptake (VO2) from baseline. Secondary endpoints will include the changes in resting and exercise-induced CBP and brachial blood pressures, number of antihypertensive medications prescribed, resting and exercise change in LV systolic and diastolic function (see below), changes in: cardiac output, exercise time, anaerobic threshold, minute ventilation (VE) over carbon dioxide produced (VCO2) slope (ventilatory efficiency). There will be a total of 7 visits, the first and last for exercise testing; the intervening 5 visits will be routine heart failure clinic follow up appointments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Cardiac Ejection Fraction (EF) greater than or equal to 25% by echocardiography within 12 months
* Stable New York Heart Association (NYHA) class II or greater
* Heart Failure consultation within the last 18 months
* Ability to exercise on a cycle ergometer
* Stable angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARB) dosage for greater than 3 months

Exclusion Criteria:

* Enrollment in a concurrent study that may confound the results of this study
* Subjects with medical conditions that would limit study participation
* Pregnancy
* Brachial Systolic Blood Pressure less than 110 mmHg
* Baseline AIx less than 15%
* Cardiac Surgery with 60 days of potential study enrollment
* Myocardial infarction within 30 days of potential study enrollment
* Hemodynamically significant valvular stenosis (greater than mild)
* Heart failure due to thyroid disease
* Active myocarditis or anemia defined as hemoglobin less than 9 mg/dl
* Presence of severe renal insufficiency with serum creatinine greater than 2.5 mg/dl
* Significant pulmonary hypertension or Cor pumonale
* Irregular heart rhythms
* Dyspnea due to pulmonary disease
* Uninterpretable echocardiographic images or radial tonometry data
* Significant competing cause for exercise intolerance (e.g., severe stable angina)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A. Borlaug, MD, Principal Investigator — Staff Physician, Mayo Clinic
Locations (2):
- United States (2):
  - University of Arizona, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Wohlfahrt P, Melenovsky V, Redfield MM, Olson TP, Lin G, Abdelmoneim SS, Hametner B, Wassertheurer S, Borlaug BA. Aortic Waveform Analysis to Individualize Treatment in Heart Failure. Circ Heart Fail. 2017 Feb;10(2):e003516. doi: 10.1161/CIRCHEARTFAILURE.116.003516. PMID 28159826
- [Derived] Borlaug BA, Olson TP, Abdelmoneim SS, Melenovsky V, Sorrell VL, Noonan K, Lin G, Redfield MM. A randomized pilot study of aortic waveform guided therapy in chronic heart failure. J Am Heart Assoc. 2014 Mar 20;3(2):e000745. doi: 10.1161/JAHA.113.000745. PMID 24650926

RESULTS

PARTICIPANT FLOW:
Groups:
- SphygmoCor Unblinded: The use of the sphygmocor values will determine medication adjustments to optimize heart failure (HF) treatment.
  SphygmoCor: The SphygmoCor, a hand-held tonometer will assess central blood pressure noninvasively. This pencil-lide device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure.
- SphygmoCor Blinded: Sphygmocor values will be blinded to the investigator.
  SphygmoCor: The SphygmoCor, a hand-held tonometer will assess central blood pressure noninvasively. This pencil-lide device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure.
Period: Overall Study
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Started | 30 | 30
Completed | 23 | 27
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Hip Surgery | 0 | 1
Not completed — Severe Peptic Ulcer Disease | 1 | 0
Not completed — Cancer | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only the participants who completed the trial were included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (8) | 72 (8) | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 16 | 23 | 39
Region of Enrollment [Number; unit: participants]
  United States | 23 | 27 | 50
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kg/m^2 | 29.2 (4.5) | 29.9 (4.6) | 29.6 (4.6)
History of Hypertension [Number; unit: participants]
  Prior Hypertension | 20 | 26 | 46
  No Prior Hypertension | 3 | 1 | 4
Diabetes [Number; unit: participants]
  Prior History of Diabetes | 12 | 12 | 24
  No History of Diabetes | 11 | 15 | 26
Obesity [Number; unit: participants]
  Obese at Baseline | 10 | 14 | 24
  Not Obese at Baseline | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake (VO2) During Maximal Effort Exercise Stress Test According to Ejection Fraction Subgroups
Description: Peak oxygen uptake (VO2) is the maximum rate of oxygen consumption as measured during incremental exercise, most typically on a motorized treadmill. Maximal oxygen consumption reflects the aerobic physical fitness of the individual. VO2 data was obtained via standard breath-by-breath expired gas analysis. Ejection Fraction Subgroups are based on participants reported at baseline.
Time Frame: baseline, 6 months
Population: For the EF subgroup 25-49%, n=48, 24 SphygmoCor Unblinded, 24 SphygmoCor Blinded. For the EF subgroup 35-49%, n=33, 14 SphygmoCor Unblinded,. 19 SphygmoCor Blinded. 2 subjects had EF either <25 or >50, and they were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change in Peak VO2
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
percentage of change in Peak VO2
  Ejection Fraction Subgroup 25-49%, n=48 | 1.5 (3.8) | -0.5 (2.5)
  Ejection Fraction Subgroup 35-49%, n=33 | 2.0 (5.4) | -1.0 (1.9)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; For 25-49% Ejection Fraction Subgroup; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; 35-49% Ejection Fraction Subgroup; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Change in Aortic Augmentation Index (AIx) According to Ejection Fraction Subgroups
Description: Aortic stiffness increases with aging, further augmenting cardiac load. One important repercussion of aortic stiffening is an increase in pulse wave velocity. As the outgoing pressure wave caused by ventricular ejection encounters zones of impedance mismatch, it is partially reflected backward, summing with the incident wave, to increase central aortic blood pressure. The magnitude of this systolic pressure wave reflection can be quantified by AIx.
  Aortic pressures were assessed in the seated position after 5 minutes rest. Aortic pulse waveform analysis was performed using a noninvasive, high-fidelity hand held tonometer placed over the radial artery. The built-in, custom software was then used to convert radial pressure waveforms to central aortic waveforms, which more accurately reflect LV afterload. The ratio of this augmented pressure to aortic pulse pressure is defined as the augmentation index (AIx).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of change in AIx
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
percentage of change in AIx
  Ejection Fraction Subgroup 25-49% | -6.9 (8.8) | -4.9 (6.3)
  Ejection Fraction Subgroup 35-49% | -8.3 (8.7) | -5.5 (6.0)

3. Secondary Outcome: Change in Heart Rate
Time Frame: baseline, six months
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
bpm | 3 (7) | -1 (10)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.06, ANOVA

4. Secondary Outcome: Change in Left Ventricle (LV) End Diastolic Volume
Description: End-diastolic volume (EDV) is the volume of blood in the right and/or left ventricle at end load or filling in (diastole). An increase in EDV increases the preload on the heart and, through the Frank-Starling mechanism of the heart, increases the amount of blood ejected from the ventricle during systole (stroke volume).
  Ventricular Data was derived from comprehensive echo-Doppler/Tissue Doppler Echo (TDE) study performed at rest, during and immediately after exercise, along with noninvasive blood pressure assessment (GE Vivid7). LV EDV was determined from the apical 4 and 2 chamber views using Simpson's method of discs, along with ejection fraction (EF).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
ml | -24 (30) | -17 (32)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.5, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Change in LV End Systolic Volume
Description: End-systolic volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole. ESV is the lowest volume of blood in the ventricle at any point in the cardiac cycle. End systolic volume can be used clinically as a measurement of the adequacy of cardiac emptying, related to systolic function.
  Ventricular Data was derived from comprehensive echo-Doppler/Tissue Doppler Echo (TDE) study performed at rest, during and immediately after exercise, along with noninvasive blood pressure assessment (GE Vivid7). LV end systolic volumes was determined from the apical 4 and 2 chamber views using Simpson's method of discs, along with EF.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
ml | -18 (18) | -11 (20)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.26, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Change in LV Ejection Fraction
Description: The ejection fraction is the percentage of the volume in the left ventricle ejected during a cardiac cycle. The normal ejection fraction is 55 to 75 percent. EF = (EDV - ESV) / EDV where EF = ejection fraction, EDV = volume of blood in the left ventricle at end-diastole, ESV = volume of blood in the left ventricle at end-systole.
  Ventricular Data was derived from comprehensive echo-Doppler/Tissue Doppler Echo (TDE) study performed at rest, during and immediately after exercise, along with noninvasive blood pressure assessment (GE Vivid7).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of LV blood volume
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
percentage of LV blood volume | 2 (2) | -0.0 (2)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.4, ANOVA

7. Secondary Outcome: Change in Stroke Volume
Description: Stroke volume (SV) is the volume of blood pumped from one ventricle of the heart with each beat. SV was determined from pulse wave (PW) and continuous wave (CW) Doppler in the LV outflow tract.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
ml | 10 (21) | 10 (21)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

8. Secondary Outcome: Change in Mitral E Velocity
Description: The Mitral E velocity is the speed at which blood fills the ventricle. It is determined by echocardiography, an ultrasound-based cardiac imaging modality.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
cm/sec | 5 (15) | 4 (12)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA

9. Secondary Outcome: Change in Mitral E/A Ratio
Description: The E/A ratio is a marker of the function of the left ventricle of the heart; it is determined by echocardiography, an ultrasound-based cardiac imaging modality. Abnormalities in the E/A ratio on Doppler echocardiography suggest that the left ventricle, which pumps blood into the circulation, cannot fill with blood properly in the period between contractions. The E/A ratio is the ratio of peak early transmitral inflow velocity and peak late mitral inflow velocity.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
ratio | -0.1 (0.3) | -0.1 (0.3)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA

10. Secondary Outcome: Change in Mitral E Wave Deceleration Time
Description: The deceleration time (DT) is the time taken from the maximum E point to baseline. Normally in adults it is less than 220 milliseconds. The DT was measured by pulse wave doppler.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- Treatment: The use of the sphygmocor values will determine medication adjustments to optimize HF treatment.
- Control: Sphygmocor values will be blinded to the investigator.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 23 | 27
milliseconds (ms) | -25 (58) | -5 (43)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.3, ANOVA

11. Secondary Outcome: Change in Brachial Systolic Blood Pressure (BP)
Description: Blood pressure is a measure of the force of the blood flowing against the walls of your arteries as it moves through your body.
  There are two numbers in a blood pressure reading. This tells how high in millimeters the pressure of your blood raises a column of mercury. The numbers usually are expressed in the form of a fraction; an example of a blood pressure reading is 120/80 mm Hg. The first, or top, number (120 in the example) is the systolic pressure. The systolic pressure is the measure of your blood pressure as the heart contracts and pumps blood. The second or lower number is the diastolic pressure and is the measure taken when your heart is at rest (80 in the example)
  Brachial systolic BP was determined by a standard oscillometric device (Dinemap, Critikon).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
mmHg | -9 (17) | -9 (24)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Test type: Superiority or Other; p = 0.24, t-test, 2 sided

12. Secondary Outcome: Change in Brachial Diastolic BP
Description: Blood pressure is a measure of the force of the blood flowing against the walls of your arteries as it moves through your body.
  There are two numbers in a blood pressure reading. This tells how high in millimeters the pressure of your blood raises a column of mercury. The numbers usually are expressed in the form of a fraction; an example of a blood pressure reading is 120/80 mm Hg. The first, or top, number (120 in the example) is the systolic pressure. The systolic pressure is the measure of your blood pressure as the heart contracts and pumps blood. The second or lower number is the diastolic pressure and is the measure taken when your heart is at rest (80 in the example)
  Brachial diastolic BP was determined by a standard oscillometric device (Dinemap, Critikon).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
mmHg | -2 (8) | -4 (14)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.6, ANOVA

13. Secondary Outcome: Change in Central Systolic BP
Description: Central blood pressure (CBP) is the pressure in the aorta, which is the large artery into which the heart pumps. This was determined by noninvasive radial tonometry, which undergoes transfer function using customized software to derive CBP tracings.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
mmHg | -8 (19) | -9 (18)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

14. Secondary Outcome: Change in Central Diastolic BP
Description: as for outcome 13
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
mmHg | -7 (10) | -3 (9)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

15. Secondary Outcome: Change in Augmentation Index
Description: as for outcome 2
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of change in AIx
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
percentage of change in AIx | -7 (9) | -5 (6)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.4, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

16. Secondary Outcome: Change in Arterial Elastance
Description: Elastance is a measure of the tendency of a hollow organ to recoil toward its original dimensions upon removal of a distending or compressing force. Effective arterial elastance was determined by the ratio of end systolic BP/stroke volume (SV).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg/ml
Arm/Group | SphygmoCor Unblinded | SphygmoCor Blinded
Number analyzed (Participants) | 23 | 27
mmHg/ml | -0.3 (0.4) | -0.3 (0.4)
Statistical Analysis 1: Comparison: SphygmoCor Unblinded vs SphygmoCor Blinded; Test type: Superiority or Other; p = 0.9, ANOVA
Statistical Analysis 2: Comparison: SphygmoCor Unblinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: SphygmoCor Blinded; Within group change compared to baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were followed for safety reporting at monthly visits over the 6-month study period.
Description: The adverse event subject population did not include the six subject who were loss to follow up, and the three subjects who withdrew because of noncardiac medical conditions that developed during the study period. Therefore adverse events are reported on 27 subjects in the control arm, and 24 subjects in the treatment arm.
Groups:
- Treatment: The use of the sphygmocor values will determine medication adjustments to optimize HF treatment.
  SphygmoCor: The SphygmoCor, a hand-held tonometer will assess central blood pressure noninvasively. This pencil-like device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure.
- Control: Sphygmocor values will be blinded to the investigator.
  SphygmoCor: The SphygmoCor, a hand-held tonometer will assess central blood pressure noninvasively. This pencil-like device is applied over the radial artery, and uses a validated mathematical transformation to derive central aortic pressure.
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 3/24 | 2/27
Other Adverse Events (participants affected / at risk) | 10/24 | 5/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24) | Control (N=27)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure Hospitalization (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=24) | Control (N=27)
Dizziness (Nervous system disorders) | 8 (8) | 5 (5)
Worsening Renal Function (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No